CLINICAL TRIAL: NCT02888301
Title: The Biodistribution of [18F]-Clofarabine in Cancer Patients Before and After Interventions That Increase the Activity of Deoxycytidine Kinase
Brief Title: 18F-Clofarabine PET/CT in Imaging Cancer Patients Before and After Interventions
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-000246; NCI-2016-00210 (Registry Identifier: CTRP); 15-000246 (Other: JCCC)
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2019-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (18F-clofarabine biodistribution): Patients receive 18F-clofarabine IV and undergo PET/CT scan at baseline and 2-4 weeks after completion of immunotherapy.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorine F 18 Clofarabine; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-clofarabine PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fluorine F 18 Clofarabine — Given IV
  Other Names: 18F-CA; 18F-Clofarabine; [18F]-Clofarabine; Cl-18F-ara-A
Procedure: Positron Emission Tomography — Undergo 18F-clofarabine PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies 18F-clofarabine positron emission tomography (PET)/computed tomography (CT) in imaging patients with cancer before and after treatment with a therapy that activates the patient's immune system (immunotherapy). PET/CT scans give detailed pictures of areas inside the body. 18F-clofarabine is a drug that contains a radioactive substance that is taken up by cells expressing deoxycytidine kinase (dCK), which is highly expressed in activated immune cells, making them light up during PET/CT scans. Doctors also want to know how 18F-clofarabine is distributed throughout the body before and after treatment with immunotherapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether positron emission tomography (PET) using the new imaging agent 18F-clofarabine can be used for imaging cancer, and whether interventions that activate the immune system can change the biodistribution of 18F-clofarabine.

OUTLINE:

Patients receive 18F-clofarabine intravenously (IV) and undergo PET/CT scan at baseline and 2-4 weeks after completion of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to tolerate PET/CT (i.e. not claustrophobic and able to remain supine)
* No restrictions based on gender or racial/ethnic background

Exclusion Criteria:

* Women of childbearing age will have to undergo a pregnancy test that will be provided free of charge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients under treatment using immune system activating interventions.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
18F-clofarabine concentration in cancer tissue | Up to 4 weeks
Change in 18F-clofarabine biodistribution | Baseline to up to 4 weeks
  For the biodistribution studies, regions of interest will be drawn on images of liver, kidney, bladder, heart, lung and blood pool to obtain regional activity count rates. Standardized uptake values (SUV = count activity per ml within region of interest (MBq-1)/(injected dose [MBq]/body weight [kgx1000]) will be calculated for different organs and for regions of tumor. Further, regional target to background count activity ratios will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Allen-Auerbach, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States